CLINICAL TRIAL: NCT01337206
Title: Evaluation of the Effectiveness of the SX ELLA Esophageal Degradable BD (BD Stent) Stent System
Brief Title: SX ELLA Esophageal Degradable BD Stent System
Acronym: DESTINY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-024
Record Dates: First submitted 2011-04-13; First posted 2011-04-18 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Benign Esophageal Lesions
Keywords: Esophageal Stenosis; Esopageal Strictures; Esophageal Dysphagia
MeSH Terms: conditions — Esophageal Stenosis; Deglutition Disorders | interventions — Stents

ARMS (2):
- Stenting Arm (Experimental): Stenting Arm
  Interventions: Device: Stenting with ELLA Biodegradable stent
- Dilation Arm (Active Comparator): Dilation Arm
  Interventions: Procedure: Standard Dilations

INTERVENTIONS:
Device: Stenting with ELLA Biodegradable stent — Treating benign esophageal lesions with the placement of a degradable stent
  Other Names: Esophageal Stenting
  Arms: Stenting Arm
Procedure: Standard Dilations — Treating benign esophageal lesions with standard dilation therapy
  Other Names: Bougie Dilation, Balloon Dilation
  Arms: Dilation Arm

SUMMARY:
The SX-ELLA Stent Esophageal Degradable BD (BD Stent) is designed for dilation of benign esophageal lesions, namely: (1) stenosis (peptic, anastomotic or caustic) refractory to standard therapy, (2) achalasia refractory to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* A recurrent benign esophageal stricture due to all causes (surgery, radiation therapy, corrosive ingestion, peptic injury, PDT, or other ablative therapy)

Exclusion Criteria:

* Patient < 18 years old
* Patient is unwilling or unable to sign and date the informed consent
* Patient is unwilling or unable to comply with the follow-up schedule
* Patient is pregnant, breast-feeding, or planning to become pregnant in the next 12 months
* Patient is simultaneously participating in another drug or device study or the patient has completed the follow-up phase for the primary objective of any previous study less than 30 days prior to enrollment in this study
* Patient with a life expectancy < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The average number of dilations per patient within 3 months / 6 months following placement of an ELLA stent | 3 - 6 months

SECONDARY OUTCOMES:
Number of patients remaining dysphagia and stricture free within 6 and 12 months after inclusion | 6 - 12 months
Time to recurrent significant dysphagia | 6 - 12 months
Time to dilation of recurrent stricture | 6 - 12 months
6 months and 12 months incidence of repeat dilation | 6 - 12 months
Serious and minor adverse events with possible or likely relation to the study Intervention | 6 - 12 months
Direct medicals costs: procedures, secondary interventions | 6 - 12 months
Quality of Life | 6 - 12 months
Technical success | 6 - 12 months
  Observing proper deployment and placement of stent using endoscopic and radiographic imaging.
Assessment of presence of gold markers within the region of the esophagus at 3 months, if possible | 6 - 12 months
  Assessment of presence of gold markers within the region of the esophagus at 3 months, using radiographic imaging, if possible, to check for remaining sections of stent that have not yet degraded.

CONTACTS AND LOCATIONS:
Overall Officials: Peter D. Siersema, MD, PhD, Principal Investigator — University Medical Center Utrech
Locations (8):
- Belgium (2):
  - Clinique Universitaire Saint Luc, Brussels
  - University Hospitals Leuven, Leuven
- IRCCS Istituto Clinico Humanitas, Milan, Italy
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - St. Antonius Hospital, Nieuwegein
  - University Medical Center Utrech, Utrecht
- Hospital General Universitario de Ciudad Real, Ciudad Real, Spain
- University College of London Hospital, London, United Kingdom

REFERENCES:
- [Derived] Walter D, van den Berg MW, Hirdes MM, Vleggaar FP, Repici A, Deprez PH, Viedma BL, Lovat LB, Weusten BL, Bisschops R, Haidry R, Ferrara E, Sanborn KJ, O'Leary EE, van Hooft JE, Siersema PD. Dilation or biodegradable stent placement for recurrent benign esophageal strictures: a randomized controlled trial. Endoscopy. 2018 Dec;50(12):1146-1155. doi: 10.1055/a-0602-4169. Epub 2018 Jun 8. PMID 29883979